CLINICAL TRIAL: NCT01249079
Title: Expanding Rapid Ascertainment Network of Schizophrenia Families in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Hsien-Yuan Lane,Chief of Psychiatry Department, China Medical University Hospital
Other Study IDs: DMR99-IRB-214
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based

GROUPS / COHORTS (1):
- Schizophrenia Family
  Interventions: Other: No intervention would be provided in this research

INTERVENTIONS:
Other: No intervention would be provided in this research — No intervention would be provided in this research,but need to draw blood

SUMMARY:
This proposal responds to Request for Applications RFA-MH-08-131, which seeks applications that propose to enrich pre-existing resources for schizophrenia in the National Institute of Mental Health (NIMH) Human Genetics Initiative and to apply genomic methods to further the investigators understanding of the molecular etiology of the disorder. The overarching aims of this proposal are to quickly and cost-effectively ascertain a large sample of trio families affected by schizophrenia, and to discover causal variants for the disorder in the first family-based genome-wide association study (GWAS) of the disorder. In Taiwan, there is no such kind of policy to support this kind of GWAS study as it is a very expensive study, including collecting large family samples and genome-wide single-nucleotide polymorphism (SNP) scanning. The investigators, thus, collaborate with Professor Ming T, Tsuang and his entended subcontracted researchers to apply for this project. The investigators, the research team in Taiwan, will collect 3800 trio families (11400 subjects) of schizophrenia. Through additional ascertainment within this framework, the investigators will collect an aggregate sample with adequate power for detecting in a GWAS those variants that make even small contributions to the risk for the disorder.

The investigators will meet the overarching goals of this project by accomplishing several Specific Aims, as follows: 1) Rapidly ascertain schizophrenia trio families from Taiwanese clinical ascertainment sites; 2) Supplement NIMH Genetics Initiative collections by sending all clinical data and biomaterials to the appropriate repositories; 3) Assess the association of schizophrenia with a genome-wide panel of single-nucleotide polymorphisms (SNPs) and their constituent haplotypes; 4) Analyze quantitative schizophrenia phenotypes such as age at onset ; 5) Perform a genome-wide survey for copy-number variations related to schizophrenia; 6) Test for gene-gene interactions (epistasis); and 7) Test for gene-environment interactions, such as the well-established effect of season of birth.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of schizophrenia and their parents, and parents are still alive

Exclusion Criteria:

* person with Mental Retardation
* persons with epilepsy
* alcohol or substance abuse combined
* in combination with other organic brain damage syndrome

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Schizophrenia patients and their biological parents
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Yuan Lane, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan